CLINICAL TRIAL: NCT01680705
Title: Ideal Frequency of Postoperative High Volume Saline Irrigations Following Endoscopic Sinus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Luke Rudmik (Other)
Responsible Party: Sponsor-Investigator, Dr. Luke Rudmik, Principal Investigator, University of Calgary
Organization: University of Calgary (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SIESS-2012
Record Dates: First submitted 2012-08-30; First posted 2012-09-07 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Rhinosinusitis
Keywords: Chronic Rhinosinusitis; Endoscopic Sinus Surgery; Sinonasal saline irrigation; Frequency; Postoperative; High Volume; Randomized Control Trial; Single Blinded; Prospective Study; Quality of Life; Endoscopic Sinus Score
MeSH Terms: conditions — Rhinosinusitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Frequency: Once Daily (Active Comparator): Patients will use high volume saline irrigation once daily post operatively.
  Interventions: Other: High Volume Saline Irrigation
- Frequency: Twice Daily (Active Comparator): Patients will use high volume saline irrigation twice daily post operatively.
  Interventions: Other: High Volume Saline Irrigation
- Frequency: Three Times Daily (Active Comparator): Patients will use high volume saline irrigation three times daily post operatively.
  Interventions: Other: High Volume Saline Irrigation

INTERVENTIONS:
Other: High Volume Saline Irrigation — High volume saline irrigation (240 ml)

SUMMARY:
The aim of this study is to determine what the ideal frequency of high-volume sinonasal saline irrigation in the early postoperative period following ESS for medically refractory CRS. We will evaluate once, twice, and three times daily frequency sinonasal saline irrigation protocols. Our hypothesis is that three times a day sinonasal saline irrigations for the first week is ideal with no difference between frequencies after 1 week.

DETAILED DESCRIPTION:
Chronic Rhinosinusitis (CRS) is a common inflammatory condition of the upper respiratory tract lasting more than 8 to 12 weeks. Major symptoms include facial congestion/fullness, facial pain/pressure, nasal obstruction/blockage, purulent nasal drainage, and reduction or loss of smell. The diagnosis must include two major symptoms and either endoscopic evidence of polyps, edema or mucopurulent discharge from the middle meatus and/or CT changes in the mucosa of sinuses or ostiomeatal complexes.

CRS has an estimated prevalence of 5% in the Canadian population, and up to 16% in some adult populations in the United States. Sinusitis is associated with a major societal health care burden, costing billions of dollars a year in North America. The medical treatment of CRS includes topical saline and corticosteroid sprays, systemic steroids and antimicrobials. Specifically, sinonasal saline irrigation is a safe, nonpharmacologic treatment, and an important and efficacious component in the management of CRS. Sinonasal saline irrigation can vary by concentration (e.g. hypertonic, isotonic, hypotonic), pressure (e.g. passive or active), and volume (e.g. high and low).

A recent evidence-based review by Rudmik et al. recommended sinonasal saline irrigation in the early postoperative period following endoscopic sinus surgery. Although 'daily' sinonasal saline irrigations are recommended, the ideal frequency is unknown since there have been no studies evaluating this topic.

This is a prospective, randomized, single blind study evaluating the subjective and objective outcomes of different sinonasal saline irrigation frequencies in patients who receive ESS for medically refractory CRS. Both disease-specific quality of life (QoL) and endoscopy scores will be measured at 1 week, 3 weeks, and 2 months postoperatively. The expected total number of patients to be enrolled in this study is approximately 75 (25 per arm), with a planned completion time of two years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a diagnosis of CRS as per guidelines (> 18 years old)
* Documented failed medical treatment of CRS
* Planned ESS for the treatment of CRS
* Able to read and understand English

Exclusion Criteria:

* Pregnant
* Cystic Fibrosis
* Diagnosed immotile cilia syndrome
* Diagnosed immunodeficiency syndrome
* Diagnosed fungal sinusitis
* Sinonasal tumours or obstructive lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life | Pre and post operative (1, 3 and 8 weeks post operatively)
  The SNOT-22 and the nasal and sinus symptoms score will be complete by the patient to assess quality of life. They will be completed preoperatively and 1 week, 3 weeks and 2 months postoperatively.

SECONDARY OUTCOMES:
Change in Endoscopic Score | Pre and Post-Operative (1, 3 and 8 weeks post operatively)
  Two endoscopic scales (the Lund-Kennedy and the POSE) will be used to assess the endoscopic appearance pre and post operatively. They will be completed preoperatively and 1 week, 3 weeks and 2 months postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Luke Rudmik, MD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Background] Desrosiers M, Evans GA, Keith PK, Wright ED, Kaplan A, Bouchard J, Ciavarella A, Doyle PW, Javer AR, Leith ES, Mukherji A, Robert Schellenberg R, Small P, Witterick IJ. Canadian clinical practice guidelines for acute and chronic rhinosinusitis. J Otolaryngol Head Neck Surg. 2011 May;40 Suppl 2:S99-193. English, French. PMID 21658337
- [Background] Chen Y, Dales R, Lin M. The epidemiology of chronic rhinosinusitis in Canadians. Laryngoscope. 2003 Jul;113(7):1199-205. doi: 10.1097/00005537-200307000-00016. PMID 12838019
- [Background] Anand VK. Epidemiology and economic impact of rhinosinusitis. Ann Otol Rhinol Laryngol Suppl. 2004 May;193:3-5. doi: 10.1177/00034894041130s502. PMID 15174752
- [Background] Ray NF, Baraniuk JN, Thamer M, Rinehart CS, Gergen PJ, Kaliner M, Josephs S, Pung YH. Healthcare expenditures for sinusitis in 1996: contributions of asthma, rhinitis, and other airway disorders. J Allergy Clin Immunol. 1999 Mar;103(3 Pt 1):408-14. doi: 10.1016/s0091-6749(99)70464-1. PMID 10069873
- [Background] Van Cauwenberge P, Watelet JB. Epidemiology of chronic rhinosinusitis. Thorax. 2000 Oct;55 Suppl 2(Suppl 2):S20-1. doi: 10.1136/thorax.55.suppl_2.s20. No abstract available. PMID 10992549
- [Background] Tomooka LT, Murphy C, Davidson TM. Clinical study and literature review of nasal irrigation. Laryngoscope. 2000 Jul;110(7):1189-93. doi: 10.1097/00005537-200007000-00023. PMID 10892694
- [Background] Rabago D, Zgierska A, Mundt M, Barrett B, Bobula J, Maberry R. Efficacy of daily hypertonic saline nasal irrigation among patients with sinusitis: a randomized controlled trial. J Fam Pract. 2002 Dec;51(12):1049-55. PMID 12540331
- [Background] Meltzer EO, Hamilos DL. Rhinosinusitis diagnosis and management for the clinician: a synopsis of recent consensus guidelines. Mayo Clin Proc. 2011 May;86(5):427-43. doi: 10.4065/mcp.2010.0392. Epub 2011 Apr 13. PMID 21490181
- [Background] Morley AD, Sharp HR. A review of sinonasal outcome scoring systems - which is best? Clin Otolaryngol. 2006 Apr;31(2):103-9. doi: 10.1111/j.1749-4486.2006.01155.x. PMID 16620328
- [Background] Wright ED, Agrawal S. Impact of perioperative systemic steroids on surgical outcomes in patients with chronic rhinosinusitis with polyposis: evaluation with the novel Perioperative Sinus Endoscopy (POSE) scoring system. Laryngoscope. 2007 Nov;117(11 Pt 2 Suppl 115):1-28. doi: 10.1097/MLG.0b013e31814842f8. PMID 18075447
- [Background] Hopkins C, Browne JP, Slack R, Lund V, Brown P. The Lund-Mackay staging system for chronic rhinosinusitis: how is it used and what does it predict? Otolaryngol Head Neck Surg. 2007 Oct;137(4):555-61. doi: 10.1016/j.otohns.2007.02.004. PMID 17903570